CLINICAL TRIAL: NCT03835598
Title: Post-Operative Thrombocytopenia After Bio-prosthesis Implantation (PORTRAIT Study): a Retrospective International Multicenter Cohort Study
Brief Title: Post-Operative Thrombocytopenia After Bio-prosthesis Implantation
Acronym: PORTRAIT
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL68980.068.19
Record Dates: First submitted 2019-02-01; First posted 2019-02-08 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-03

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cardiac biological prosthesis

SUMMARY:
The objective of the study is to obtain the clinical data from patients who received a biological prosthesis in aortic or mitral position, in order to evaluate the occurrence of peri-operative thrombocytopenia.

The aim of the study is to analyze the eventual clinical impact of the phenomenon (re-operation for bleeding, blood transfusion) and the mortality rate.

This is a multicentre retrospective, observentional clinical study. This study will enroll up to 5000 patients since 2000 to date.

DETAILED DESCRIPTION:
Cardiac surgery is commonly associated with a transient post-operative decrease in the platelet count. Thrombocytopenia after cardiopulmonary bypass can be explained by hemodilution, exposure to artificial surfaces with platelet activation and adhesion, hypothermia, blood loss and mechanical sequestration. It usually occurs between the second and third postoperative days, resulting in a reduction of platelet counts by 40-50% from baseline values. Moreover, when a foreign body as a valve prosthesis is literally placed into the blood flow, blood cells are constantly exposed to its surface and eventually inflammatory and, perhaps, autoimmune reactions could start. The interactions biomaterial-blood induce changes in platelet shape, metabolism as well as receptor-mediated dysfunction and lysis. Then, any significant decline in the circulating platelet count raises concerns about coagulation disorders and bleeding.

Despite the advanced hemodynamic performance, recently thrombocytopenia (defined as nadir platelet count < 150.000 x 1000/uL) has been associated to new aortic biological prostheses, either rapid deployment or trans-catheter valves. Although several studies have been carried on, the drop in the platelet count after aortic valve replacement with certain tissue valves remains unexplained yet. The decrease after the valve implantation, however, is not exclusively limited to the surgical prostheses. Trans-catheter aortic valves, in fact, were found to be associated to post-procedure thrombocytopenia. Thrombocytopenia following transcatheter aortic valve implantation (TAVI) procedures is related to the increased adverse events rate such as death, stroke, acute kidney injury, bleeding and vascular complications. Furthermore, thrombocytopenia seems to occur most likely associated after balloon-expandable valves implantation.The literature, however, is confounding.

Despite several studies, little is known about the mechanism involved. Variations in biocompatibility of valve tissue as like a strong immune/inflammatory response could be some explanations. However, there is still uncertainty about the mechanism conditioning post-operative platelet drop. To address this uncertain the underlying process should be evaluated in a large multicentre trial.

The aims of the study are the following:

* to analyze the occurrence of thrombocytopenia after isolated aortic valve replacement/implantation and after isolated mitral valve replacement;
* to evaluate the clinical impact of thrombocytopenia (length of stay, bleeding, re-operation for bleeding, blood transfusion, mortality).

The study is multicentre, retrospective, observational and will enroll up to 5000 since 2000 to date.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated aortic valve replacement/implantation or isolated mitral valve replacement with a biological prosthesis.

Exclusion Criteria:

* Pre-existent thrombocytopenia;
* Oncologic diseases;
* Pre-existent infections/inflammations;
* Use of drugs inducing thrombocytopenia (<3months);
* Combined cardiac surgery operations;
* Recent percutaneous cardiac intervention (<1month).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is composed by adult patients submitted to isolated aortic valve replacement, percutaneous trans-catheter aortic valve implantation, and mitral valve replacement with a bio-prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 1233 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Platelet count | During the index hospital stay, an average of 5 days
  to evaluate the rate of thrombocytopenia in patients receiving biological prosthesis
Platelet count | 1-3months follow-up
  to evaluate the rate of thrombocytopenia in patients receiving biological prosthesis
packed Red Cells transfusion, fresh frozen plasma transfusion, Platelet transfusion | During the index hospital stay, an average of 5 days
  to determine the low platelets-related complication rate
Major bleeding (requiring more than 2 Red blood cells transfusions) | From the index procedure up to 3 months
  to determine the low platelets-related complication rate
Re-exploration for bleeding | From the index procedure up to 3 months
  to determine the low platelets-related complication rate

SECONDARY OUTCOMES:
In-hospital mortality | Participants are followed during the duration of hospital stay (expected: up to 7 days post-op)
  to assess the in-hospital mortality
In-hospital length of stay | From the index procedure through discharge from the hospital (expected: up to 7 days post-op)
  Days after the prosthesis implantation
ICU length of stay | From the index procedure through discharge from the Intensive Care Unit (expected: up to 2 days post op)
  Days after the prosthesis implantation
Gastro-intestinal bleeding | From the index procedure within 3 months
  Occurrence of gastro-intestinal bleeding
Intracranial Bleeding | From the index procedure within 3 months
  Occurrence of intra-cranial bleeding
Thrombosis | From the index procedure within 3 months
  Occurrence of Thrombosis (arterial or venous)
30-day mortality | within 30 days
  Mortality within 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Federica Jiritano, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yerebakan C, Kaminski A, Westphal B, Kundt G, Ugurlucan M, Steinhoff G, Liebold A. Thrombocytopenia after aortic valve replacement with the Freedom Solo stentless bioprosthesis. Interact Cardiovasc Thorac Surg. 2008 Aug;7(4):616-20. doi: 10.1510/icvts.2007.169326. Epub 2008 May 27. PMID 18505752
- [Background] Reents W, Babin-Ebell J, Zacher M, Diegeler A. Thrombocytopenia after aortic valve replacement with the Sorin Freedom Solo prosthesis. J Heart Valve Dis. 2011 May;20(3):313-8. PMID 21714423
- [Background] Repossini A, Tononi L, Martinil G, Di Bacco L, Girolettiz L, Rosati F, Muneretto C. Platelet activation after sorin freedom solo valve implantation: a comparative study with Carpentier-Edwards Perimount Magna. J Heart Valve Dis. 2014 Nov;23(6):777-82. PMID 25790627
- [Background] Albacker TB. Thrombocytopenia associated with Perceval sutureless aortic valve replacement in elderly patients: a word of caution. Heart Surg Forum. 2015 Jun 26;18(3):E093-7. doi: 10.1532/hsf.1324. PMID 26115151
- [Background] Stanger O, Grabherr M, Gahl B, Longnus S, Meinitzer A, Fiedler M, Tevaearai H, Carrel T. Thrombocytopaenia after aortic valve replacement with stented, stentless and sutureless bioprostheses. Eur J Cardiothorac Surg. 2017 Feb 1;51(2):340-346. doi: 10.1093/ejcts/ezw295. No abstract available. PMID 28186236
- [Background] Gallet R, Seemann A, Yamamoto M, Hayat D, Mouillet G, Monin JL, Gueret P, Couetil JP, Dubois-Rande JL, Teiger E, Lim P. Effect of transcatheter (via femoral artery) aortic valve implantation on the platelet count and its consequences. Am J Cardiol. 2013 Jun 1;111(11):1619-24. doi: 10.1016/j.amjcard.2013.01.332. Epub 2013 Mar 20. PMID 23523059
- [Background] Jilaihawi H, Doctor N, Chakravarty T, Kashif M, Mirocha J, Cheng W, Lill M, Nakamura M, Gheorghiu M, Makkar RR. Major thrombocytopenia after balloon-expandable transcatheter aortic valve replacement: prognostic implications and comparison to surgical aortic valve replacement. Catheter Cardiovasc Interv. 2015 Jan 1;85(1):130-7. doi: 10.1002/ccd.25430. Epub 2014 Feb 27. PMID 24677617